CLINICAL TRIAL: NCT04272216
Title: The RAVI Registry: A Prospective, Multi-Center, Observational Study of Radial Access Embolization Procedures Using HydroPearl Microspheres
Brief Title: An Observational Study of Radial Access Embolization Procedures Using HydroPearl Microspheres
Acronym: RAVI Registry
Status: Completed | Type: Observational
Sponsor: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TIS2019-02
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2021-10

CONDITIONS: Uterine Fibroid; Arteriovenous Malformations; Hypervascular Tumors; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Leiomyoma; Arteriovenous Malformations; Prostatic Hyperplasia | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Treatment with HydroPearl via radial access: all patients will be in the same group/cohort in this open-label, single-arm, observational registry.
  Interventions: Device: Treatment with HydroPearl via radial access

INTERVENTIONS:
Device: Treatment with HydroPearl via radial access — This is an observational study collecting data on patients who are already being treated with HydroPearl on-label per standard of care.

SUMMARY:
This registry study is designed to collect data on the procedural success and complication rates in real-world patients undergoing HydroPearl embolization procedures via radial access.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old
2. Subject is scheduled for a procedure for treatment with HydroPearl microspheres using radial access.
3. Subject is willing and able to complete follow-up requirements
4. Subject is willing and able to sign a written Informed Consent form prior to participating in the registry.

Exclusion Criteria:

1. Unable to have a procedure with radial access for any reason.
2. Participating in another clinical study which, in the opinion of the investigator, could impact the results of this registry.
3. Pregnant or planning to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multi-center, registry study to assess the procedural success, technical success, and complication rate of radial access procedures using HydroPearl microspheres.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2023-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Guimaraes, MD, Principal Investigator — Medical University of South Carolina
Locations (6):
- United States (6):
  - University of California - Los Angeles, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - SLU Department of Radiology, St Louis, Missouri
  - Mount Sinai, New York, New York
  - UNC, Chapel Hill, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Uterine Fibroid Embolization With HydroPearls Via Radial Access: Patients will be separated into the following groups based on indication:
  Uterine Fibroid Embolization (UFE)
  All subjects will receive treatment with HydroPearl via radial access.
- Prostatic Artery Embolization With HydroPearls Via Radial Access: Patients will be separated into the following groups based on indication:
  Prostatic Artery Embolization (PAE) to treat benign prostatic hyperplasia (BPH).
  All subjects will receive treatment with HydroPearls via radial access.
- Liver Tumor Embolization With HydroPearls Via Radial Access: Patients will be separated into the following groups based on indication:
  Liver Tumor Embolization (LT) to hypervascular tumors in the liver.
  All subjects will receive treatment with HydroPearls via radial access.
- Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access: Patients will be separated into the following groups based on indication:
  Other Hypervascular Tumors (OHT) to treat hypervascular tumors located outside of the liver.
  All subjects will receive treatment with HydroPearls via radial access.
Period: Overall Study
Arm/Group | Uterine Fibroid Embolization With HydroPearls Via Radial Access | Prostatic Artery Embolization With HydroPearls Via Radial Access | Liver Tumor Embolization With HydroPearls Via Radial Access | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access
Started | 70 | 16 | 7 | 6
Completed | 45 | 8 | 2 | 5
Not Completed | 25 | 8 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uterine Fibroid Embolization With HydroPearls Via Radial Access | Prostatic Artery Embolization With HydroPearls Via Radial Access | Liver Tumor Embolization With HydroPearls Via Radial Access | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access | Total
Number analyzed (Participants) | 70 | 16 | 7 | 6 | 99
Age, Continuous [Mean (Full Range); unit: years] | 44.3 [32.0 to 54.0] | 67.6 [55 to 82.0] | 59.6 [40 to 66] | 60.3 [49 to 68] | 50.1 [32 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 0 | 1 | 3 | 74
  Male | 0 | 16 | 6 | 3 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 44 | 1 | 3 | 1 | 49
  White | 19 | 14 | 4 | 5 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 70 | 16 | 7 | 6 | 99
Medical History [Count of Participants; unit: Participants]
  Myocardial Infarction (MI) | 1 | 1 | 0 | 0 | 2
  Atrial Fibrillation | 0 | 4 | 0 | 0 | 4
  Hypertension | 26 | 7 | 4 | 6 | 43
  Hypercholesterolemia | 3 | 4 | 1 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Procedural Success
Description: Defined as completing the planned procedure without femoral access bailout
Time Frame: Duration of procedure (measured from the time the participant is sedated (start of study procedure) until all products are removed from the participant and closure is confirmed (end of the intended study procedure))
Measure: Count of Participants; unit: Participants
Arm/Group | Uterine Fibroid Embolization With HydroPearls Via Radial Access | Prostatic Artery Embolization With HydroPearls Via Radial Access | Liver Tumor Embolization With HydroPearls Via Radial Access | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access
Number analyzed (Participants) | 70 | 16 | 7 | 6
Participants | 70 | 16 | 7 | 6

2. Primary Outcome: Technical Success
Description: Delivery of HydroPearls to the target vessel and slowing the blood flow with microsphere embolization
Time Frame: Duration of procedure (from when the injection of HydroPearls is started until access site closure has been completed)
Measure: Count of Participants; unit: Participants
Arm/Group | Uterine Fibroid Embolization With HydroPearls Via Radial Access | Prostatic Artery Embolization With HydroPearls Via Radial Access | Liver Tumor Embolization With HydroPearls Via Radial Access | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access
Number analyzed (Participants) | 70 | 16 | 7 | 6
Participants
  Successful delivery of HydroPearls to target vessels | 69 | 16 | 7 | 6
  Complete Embolization | 69 | 14 | 7 | 6
  Partial Embolization | 1 | 2 | 0 | 0

3. Primary Outcome: Freedom From Major Adverse Events and Radial Access Complications
Description: Major Adverse Events are defined as the following:
  Death MI Stroke
Time Frame: within 30 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Uterine Fibroid Embolization With HydroPearls Via Radial Access | Prostatic Artery Embolization With HydroPearls Via Radial Access | Liver Tumor Embolization With HydroPearls Via Radial Access | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access
Number analyzed (Participants) | 70 | 16 | 7 | 6
Participants
  Freedom from Major Adverse Events and radial access complications within 30 days post procedure | 69 | 16 | 6 | 6
  Death within 30 days | 1 | 0 | 1 | 0
  MI within 30 days | 0 | 0 | 0 | 0
  Stroke within 30 days | 0 | 0 | 0 | 0

4. Primary Outcome: Radial Access Related Complications Within 30 Days
Description: Radial access related complications that occurred within 30 days of the index procedure include, but are not limited to, the following:
  Radial Artery Occlusion (RAO) Hand Ischemia Arteriovenous Fistula Pseudoaneurysm Any complication requiring surgical and/or endovascular intervention within 30 days of the index procedure
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Uterine Fibroid Embolization With HydroPearls Via Radial Access | Prostatic Artery Embolization With HydroPearls Via Radial Access | Liver Tumor Embolization With HydroPearls Via Radial Access | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access
Number analyzed (Participants) | 70 | 16 | 7 | 6
Participants
  Vessel occlusion | 0 | 0 | 0 | 0
  Hand Ischemia | 0 | 0 | 0 | 0
  Arteriovenous fistula | 0 | 0 | 0 | 0
  Pseudoaneurysm | 0 | 0 | 0 | 0
  Vessel dissection | 0 | 0 | 0 | 0
  Vessel spasm | 4 | 0 | 1 | 1
  Artery perforation | 0 | 0 | 0 | 0
  Distal embolization | 0 | 0 | 0 | 0
  Hematoma at the puncture site | 4 | 2 | 1 | 1
  Access site pain | 0 | 0 | 0 | 1
  Finger amputation/ loss of limb | 0 | 0 | 0 | 0
  Other | 8 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Within 30 days of index procedure
Arm/Group | Uterine Fibroid Embolization With HydroPearls Via Radial Access | Prostatic Artery Embolization With HydroPearls Via Radial Access | Liver Tumor Embolization With HydroPearls Via Radial Access | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access
All-Cause Mortality (participants affected / at risk) | 1/70 | 0/16 | 1/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/70 | 0/16 | 1/7 | 2/6
Other Adverse Events (participants affected / at risk) | 32/70 | 9/16 | 4/7 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uterine Fibroid Embolization With HydroPearls Via Radial Access (N=70) | Prostatic Artery Embolization With HydroPearls Via Radial Access (N=16) | Liver Tumor Embolization With HydroPearls Via Radial Access (N=7) | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access (N=6)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Acute hypoxic respiratory failure - not related to technique or device
Death (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — End stage liver disease - not related to procedure or device
Blood loss anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona Virus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uterine Fibroid Embolization With HydroPearls Via Radial Access (N=70) | Prostatic Artery Embolization With HydroPearls Via Radial Access (N=16) | Liver Tumor Embolization With HydroPearls Via Radial Access (N=7) | Other Hypervascular Tumor Embolization With HydroPearls Via Radial Access (N=6)
Abdominal Pain (Gastrointestinal disorders) | 11 (11) | 0 (0) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (7) | 1 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vascular access site bruising (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Genital paraesthesia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal hematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arterial Spasm (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Post embolization syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasospasm (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04272216/Prot_SAP_000.pdf